CLINICAL TRIAL: NCT03411434
Title: Added Value of the Oculomotor and Cognitive Examination in the Management of Patients With Attention Deficit Disorder With or Without Hyperactivity. Interventional Study to Evaluate Current Care
Brief Title: Added Value of the Oculomotor and Cognitive Examination in the Management of Patients With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Rouffach (Other)
Responsible Party: Principal Investigator, Fabrice Duval, MD, Psychiatrist, Centre Hospitalier Rouffach
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AO-005/20131104
Record Dates: First submitted 2018-01-12; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: oculomotor performances; neurocognition; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Interventional study designed to evaluate routine care. The patients are their own controls. Oculomotor and neurocognitive performances are assessed at baseline (V0), during the methylphenidate test (V1), and after 6 months of methylphenidate treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADHD patients (Experimental): 90 patients will be enrolled and assessed (i.e., neurocognitive and oculomotor tests) at baseline ; after a single low dose of methylphenidate (10 mg orally); and after 6 months of adequate dose of methylphenidate oral tablet
  Interventions: Drug: Methylphenidate Oral Tablet

INTERVENTIONS:
Drug: Methylphenidate Oral Tablet — cf arm group description
  Other Names: oculometry (eye tracking); neurocognition (TAP battery)

SUMMARY:
ADHD is a neurodevelopmental disorder characterized by symptoms of inattention and / or hyperactivity-impulsivity that affects nearly 6% of school-aged children and persists into adulthood. More and more studies are interested in biomarkers of this pathology. The oculomotricity, which allows to highlight deficits motor and attention present in ADHD, is used routinely in the expert centers. In general, the pharmacological treatment of ADHD is associated with a clinical response in approximately 70% of cases. Today, there is no review to predict the individual response to treatment.

Hypotheses The investigators hypothesize that a precise analysis of the oculomotor markers will allow to measure the improvement of the symptomatology of the ADHD disorder following the introduction of the psycho-stimulatory treatment. In other words, the investigators hypothesize that these markers could be a useful aid in patient follow-up by the clinician and allow early identification of responder and non-responder patients.

Primary objective The main objective of this study is to measure the added value of oculomotor examination in the follow-up of psycho-stimulant-treated ADHD patients.

Main Evaluation Criteria The primary endpoint is oculomotor performance. Parameters analyzed for each saccade are latency, amplitude, duration, average speed, direction.

Secondary Criteria Evaluation (s) Correlations will be established between oculomotor data and scores obtained at the clinical scales assessing ADHD symptoms of inattention and hyperactivity as well as cognitive performance. The data obtained before the introduction of the psycho-stimulant treatment (V0, baseline) will be compared with those obtained after acute administration of methylphenidate (10 mg orally,V1) and during the follow-up visit at 6 months (V2).

DETAILED DESCRIPTION:
Type of study and experimental plan:

This is an interventional study designed to evaluate routine care. Number of Necessary Subjects Participants will be stratified by age to control the effect of age. The age groups to be analyzed are: 7-9 vs 10-12 vs. 13-18 versus 19-29 vs 30-40 and 41-50, each with at least 15 participants. total of 90 participants.

• Study population The patients included in this study are followed in the general psychiatric department of the Rouffach hospital center for attention deficit disorder with or without hyperactivity (ADHD). The study focuses on ADHD patients aged 7 to 50 years, undergoing an oculomotor and cognitive examination before the initiation of psychostimulant therapy with methylphenidate (MPH) (baseline, V0); two weeks later (V1) following a single low dose administration of MPH (10 mg orally given at 8 AM) ; and at 6-month follow-up (V2) when patients are medicated with adequate dose of MPH.

• Clinical assessments All subjects are evaluated directly by psychiatrists and neuropsychologists who are experts in the field of ADHD and are experienced in the use of standardized or semi-standardized clinical instruments. Clinical investigation allows extensive and standardized evaluation of patients.

1. Categorical standardized assessment of ADHD symptoms Diagnostic and Statistical Manual (DSM-IV-TR) ADHD Criteria: Subtype: Combined, Inattentive, Hyperactive-Impulsive.

   • In children-adolescents: CONNERS Evaluation Scale for Teachers and Parents: Hetero-Questionnaire for Assessing Behavioral Disorders in ADHD.

   ADHD Questionnaire: self-assessment questionnaire for children and adolescents with attention difficulties, agitation and behavioral problems allowing the quantification of ADHD symptoms.

   ADHD Questionnaire: Hetero-evaluation questionnaire for children and adolescents with attention difficulties, agitation and behavioral problems allowing the quantification of ADHD symptoms. This questionnaire is completed by one of the parents.

   • In adults: Adult Self Reporting Scale (ASRS 1.1): self-assessment grid to assess current adult ADHD disorders.

   Diagnostic Interview for ADHD in adults (DIVA 2.0): semi-structured interview corresponding to the DSM-IV criteria, according to which the diagnosis of ADHD in adults requires the demonstration of symptoms of ADHD both in childhood and at age adult. This scale is composed of 3 parts that apply each to childhood and adulthood: inattention criteria, hyperactivity-impulsivity criteria, age of onset and impaired functioning due to symptoms.

   Wender Utah Rating Scale (WURS-25): a self-report scale that allows retrospective assessment of the presence of ADHD registry disorders in childhood.

   World Health Organization Disability Assessment Schedule (WHODAS 2.0): Self-Assessment Scale, to measure pathology-induced disability in daily living during the last 30 days.
2. Standardized neurocognitive assessment

   * Intellectual level The intellectual level of the patients is assessed using the Wechsler scales: Wechsler Preschool and Primary Scale of Intelligence (WIPPSI) and Wechsler Intelligence Scale for Children (WISC-IV) according to the age of the subject. The variety of tests proposed by the Wechsler Ladders allows to appreciate the level of cognitive development of the child and adolescents. Adults benefit from Adaptation French National Adult Reading Scale (fNART) which aims to estimate the intellectual pre-morbid level. It consists of a series of 40 words of the French language. The patient is asked to read each word aloud whether or not they know the word. It is therefore necessary to deduce the pronunciation of the word in question.
   * Computerized neurocognitive tests o In children up to 10 years

   KITAP computerized battery: 6 tests of this battery have been selected and are administered in the following order:
   * alert
   * divided attention
   * flexibility
   * go no go
   * distractibility
   * sustained attention o In children from 11 years old/teenagers/adults

   Computer Battery TAP 2.2: 8 tests of this battery have been selected and are administered in the following order:
   * phasic attention
   * divided attention
   * flexibility
   * incompatibility
   * go no go
   * visual scan
   * working memory
   * sustained attention The total pass of these tests lasts approximately 45 minutes to which are added 5 minutes of explanation and test (s) for each task (5 x 8). Total duration of the TAP battery run: approximately 1h25.

     • Other neurocognitive tests

     o In children:
   * Memory test
   * 15 words of Rey
   * Memory test - figures
   * Dam tests
3. Standardized assessment of psychiatric comorbidities other than ADHD

   - In children-adolescents: Social Communication Questionnaire S.C.Q - Social Communication Questionnaire): A tool for identifying the manifestations of Autonomic Spectrum Disorders in three main functional areas: social relations, communication and restricted, stereotyped and repetitive behaviors. Hetero-quiz for parents or a person who knows the child well.

   C.A.S.T The Childhood Asperger Syndrome Test: hetero-questionnaire to assess the manifestations of Asperger syndrome.

   - In adults: Semi-structured psychiatric interview. Questionnaire Mood Disorder Questionnaire (MDQ): self-questionnaire "mood disorders" allowing screening for bipolar disorders
4. Standardized evaluation of oculomotor behavior Visually guided horizontal and vertical saccade tests: A fixation point is shown in the center of the screen, after a time interval of 200 ms, the center point disappears and a new point appears on the right or left at 20 ° from the initial position. The eyes must move on the new target. Thirty horizontal and 30 vertical saccades are presented Voluntary horizontal saccadic tests: The parameters are identical to those exposed in visually guided saccadic tests except that the central point does not disappear when the second point appears on the right or on the left (top or bottom) at 20 ° from the central point. Thirty horizontal saccades are presented.

   Anti-saccadic tests: A fixation point is presented in the center of the screen, after an interval of 200ms, the central point disappears and a new point appears on the right or on the left (top or bottom) at 20 ° from the initial position. The eyes must be pointing away from the point. Thirty horizontal saccades are presented.

   All oculomotor tests last 1 minute. Horizontal and vertical chase tests: A target moves on the screen for about 50 seconds, the eyes must follow the target. The speed of the target varies from 5 ° Reading and Visual Search Tests: A text of 4 lines is presented on the computer screen. The participants must read it in a low voice, the movements of the eyes are recorded while they perform the task.

   In the visual search test, the same text is presented but all vowels are replaced by consonants. Participants must count in low voices the number of 'r' present in the text.
5. Other parameters collected Sociodemographic data, personal and family psychiatric and somatic antecedents as well as previous and current treatments are collected.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis according to DSM-IV-TR criteria
* Beneficiary of a social security scheme
* Having undergone an oculomotor examination as part of their usual care
* Normal neurological examination

Exclusion Criteria:

* Intellectual Disability (IQ < 70)
* Proven neurological pathology or identified genetic syndrome
* Vestibular pathology
* Ear, nose, and throat (ENT) pathology
* Neuro-ophthalmological pathology uncorrected by corrective glass (<10/10 in binocular vision

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-02-17 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in saccade latency after acute and chronic 6-month administration of methylphenidate vs. baseline | Baseline (V0); methylphenidate test (V1; i.e., two weeks after V0, one hour after ingestion of a single low dose administration of MPH [10 mg orally given at 8 AM]); after 6 month's treatment with methylphenidate oral tablet (V2)
  Latency (time between the onset of the target and the beginning of the eye movements in milliseconds)
Change in saccade average speed after acute and chronic 6-month administration of methylphenidate vs. baseline | Baseline (V0); methylphenidate test (V1; i.e., two weeks after V0, one hour after ingestion of a single low dose administration of MPH [10 mg orally given at 8 AM]); after 6 month's treatment with methylphenidate oral tablet (V2)
  Average speed of the saccade (degree per second)
Change in saccade accuracy after acute and chronic 6-month administration of methylphenidate vs. baseline | Baseline (V0); methylphenidate test (V1; i.e., two weeks after V0, one hour after ingestion of a single low dose administration of MPH [10 mg orally given at 8 AM]); after 6 month's treatment with methylphenidate oral tablet (V2)
  Saccade accuracy (characterized by the ratio of the amplitude of the first saccade to the amplitude of the target, expressed in percentage)
Change in direction errors after acute and chronic 6-month administration of methylphenidate vs. baseline | Baseline (V0); methylphenidate test (V1; i.e., two weeks after V0, one hour after ingestion of a single low dose administration of MPH [10 mg orally given at 8 AM]); after 6 month's treatment with methylphenidate oral tablet (V2)
  Direction errors (in percentage)
Change in anticipatory saccades after acute and chronic 6-month administration of methylphenidate vs. baseline | Baseline (V0); methylphenidate test (V1; i.e., two weeks after V0, one hour after ingestion of a single low dose administration of MPH [10 mg orally given at 8 AM]); after 6 month's treatment with methylphenidate oral tablet (V2)
  Anticipatory saccades (saccade initiated < 80 msec after target appearance, in percentage)
Change in express saccades after acute and chronic 6-month administration of methylphenidate vs. baseline | Baseline (V0); methylphenidate test (V1; i.e., two weeks after V0, one hour after ingestion of a single low dose administration of MPH [10 mg orally given at 8 AM]); after 6 month's treatment with methylphenidate oral tablet (V2)
  Express saccades (reaction time between 80 and 130 msec, expressed in percentage).

SECONDARY OUTCOMES:
Associations between clinical outcome after 6 month's methylphenidate treatment and change in oculomotor performance (from V0 to V1, V0 to V2, and V1 to V2) | Baseline (V0); methylphenidate test (V1; i.e., two weeks after V0, one hour after ingestion of a single low dose administration of MPH [10 mg orally given at 8 AM]); after 6 month's treatment with methylphenidate oral tablet (V2)
  Clinical Global Impression (CGI). The CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). Global improvement or change (CGI-C) scores range from 1 (very much improved) through to 7 (very much worse). Treatment response ratings should take account of both therapeutic efficacy and treatment-related adverse events and range from 0 (marked improvement and no side-effects) and 4 (unchanged or worse and side-effects outweigh the thera- peutic effects). Each component of the CGI is rated separately; the instrument does not yield a global score.
Associations between oculomotor data and neurocognitive test results | Baseline (V0); methylphenidate test (V1; i.e., two weeks after V0, one hour after ingestion of a single low dose administration of MPH [10 mg orally given at 8 AM]); after 6 month's treatment with methylphenidate oral tablet (V2)
  computerized neurocognitive tests (KITAP for children up to 10 years; TAP for children above 11 years, adolescents, and adults)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Duval, Principal Investigator — Centre Hospitalier Rouffach
Locations (1):
- Centre Hospitalier Rouffach, Rouffach, Alsace, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munoz DP, Armstrong IT, Hampton KA, Moore KD. Altered control of visual fixation and saccadic eye movements in attention-deficit hyperactivity disorder. J Neurophysiol. 2003 Jul;90(1):503-14. doi: 10.1152/jn.00192.2003. Epub 2003 Apr 2. PMID 12672781
- [Background] Kurscheidt JC, Peiler P, Behnken A, Abel S, Pedersen A, Suslow T, Deckert J. Acute effects of methylphenidate on neuropsychological parameters in adults with ADHD: possible relevance for therapy. J Neural Transm (Vienna). 2008;115(2):357-62. doi: 10.1007/s00702-008-0871-4. Epub 2008 Feb 12. PMID 18264813
- [Derived] Duval F, Erb A, Mokrani MC, Weiss T, Carcangiu R. First-Dose Methylphenidate-Induced Changes in the Anti-Saccade Task Performance and Outcome in Adults with Attention-Deficit/Hyperactivity Disorder. Psychiatr Res Clin Pract. 2021 May 19;3(4):146-152. doi: 10.1176/appi.prcp.20210010. eCollection 2021 Winter. PMID 36101656